CLINICAL TRIAL: NCT00697619
Title: A Prospective, Open-label, Randomized Phase III Study to Evaluate the Efficacy of ZOMETA® (Zoledronic Acid) in Treatment of Bone Metastases in Patients With Stage IV Nasopharyngeal Cancer
Brief Title: To Evaluate the Efficacy of ZOMETA® in Treatment of Bone Metastases in Patients With Stage IV Nasopharyngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Li Zhang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446ECN02
Record Dates: First submitted 2008-06-11; First posted 2008-06-16 (Estimated); Results first posted 2012-03-02 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2011-12

CONDITIONS: Nasopharyngeal Cancer
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Group (Experimental): Zometa (zoledronic acid) 4 mg over 15 min IV infusion, every 4 week Anti-neoplastic therapy .Patients can receive concomitant cycles of chemotherapy or radiotherapy.
  Interventions: Drug: Zometa (zoledronic acid)
- Contorl Group (No Intervention): Anti-neoplastic therapy alone. Patients can receive concomitant cycles of chemotherapy or radiotherapy.

INTERVENTIONS:
Drug: Zometa (zoledronic acid) — Zometa 4 mg IV infusion every 4 weeks for 24 months. Co-administration with Zometa: Calcium 500 mg + vitamin D 400-500 IU daily
  Other Names: Zometa
  Arms: Test Group

SUMMARY:
The purpose of this study is to assess the efficacy of addition of zometa to anti-neoplastic treatment compared with anti-neoplastic treatment alone, as measured by the primary efficacy variable of SREs (Skeletal Related Events) and to assess the safety in nasopharyngeal patients with bone metastases randomized to receive either zometa 4 mg or anti-neoplastic treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Age >18, either sex
* Histologically confirmed stage IV nasopharyngeal cancer
* One bone metastasis at least confirmed by imaging
* without chemotherapy or radiotherapy after bone metastasis
* Life expectancy > 6 M
* ECOG <= 2
* Adequate bone marrow reserve (WBC > 3.5 x 109/L, Neutrophile > 1.5 x 109/L, Platelet 100 x 109/L, Hb > 90 g/L)
* Serum creatinine< 2.0 mg/dL (< 1.5 times the upper limit of the normal range for the laboratory of the study center)
* Signed ICF

Exclusion Criteria:

* Women who are pregnant or in lactation
* Patients with hyperostosis
* Systemic treatment for another cancer within the year prior to study entry
* Previous or current treatment with any other bisphosphonates, bone- protecting, cytotoxic or targeted therapy
* Initial serum creatinine >265 micromol/L and/or progressive renal disease
* Known hypersensitivity to any of the study drugs or to drugs with similar chemical structures
* Use of investigational agents within 28 days of the Baseline visit, or participating simultaneously in any other clinical studies
* Severe co-morbidity of any type that may interfere with assessment of the patient for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-09; Primary Completion 2009-01 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Master, Principal Investigator — Cancer Center of Sun Yat-Sen University (CCSU)
Locations (1):
- Li Zhang, Guangzhou, Guangdong, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Anti-neoplastic therapy alone. Patients can receive concomitant cycles of chemotherapy or radiotherapy.
Period: Overall Study
Arm/Group | Test Group | Control Group
Started | 30 | 30
Completed | 24 | 22
Not Completed | 6 | 8
Not completed — Lack of Efficacy | 2 | 2
Not completed — Adverse Event | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Group | Control Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 29 | 59
  >=65 years | 0 | 1 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 46 (10) | 41 (11) | 44 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 25 | 27 | 52
Region of Enrollment [Number; unit: participants]
  China | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Comparing the Level of Urinary N-telopeptide (uNTx) in the Two Arms .
Time Frame: Baseline, the first, second and third month
Measure: Median (Standard Error); unit: nM /mM
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 30 | 29
nM /mM
  Baseline | 75 (15) | 94 (16)
  the first month | 29 (12) | 88 (23)
  the second month | 17 (7) | 52 (21)
  the third month | 11 (20) | 45 (27)
Statistical Analysis 1: Comparison: Test Group vs Control Group; Test type: Superiority or Other; p = 0.370, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Test Group vs Control Group; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Test Group vs Control Group; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Test Group | Control Group
Serious Adverse Events (participants affected / at risk) | 15/30 | 17/29
Other Adverse Events (participants affected / at risk) | 15/30 | 16/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Group (N=30) | Control Group (N=29)
Leukopenia (Blood and lymphatic system disorders) | 13 | 13
Neutropenia (Blood and lymphatic system disorders) | 8 | 7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test Group (N=30) | Control Group (N=29)
bone pain, nausea, anemia, vomiting,constipation, dyspnea and fatigue (General disorders) | 15 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No